CLINICAL TRIAL: NCT00319332
Title: A Multi-center, Randomized, Phase 3 Study of Iodine I 131 Tositumomab Therapeutic Regimen Versus Ibritumomab Tiuxetan Therapeutic Regimen for Patients With Relapsed or Transformed Follicular Non-Hodgkin's Lymphoma
Brief Title: A Comparative Study Of Iodine I 131 Tositumomab Therapeutic Regimen Versus Ibritumomab Tiuxetan Therapeutic Regimen
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study has been cancelled prior to enrollment
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 393229/029; CCBX001-053; NCT00078676 (obsolete NCT alias)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Lymphoma, Small Cleaved-Cell, Follicular; Lymphoma, Large-Cell, Follicular; Lymphoma, Follicular; Lymphoma, Non-Hodgkin
Keywords: non-Hodgkin's Lymphoma; follicular lymphoma; BEXXAR; ZEVALIN; Iodine I 131 Tositumomab; Ibritumomab Tiuxetan; Follicular, mixed small-cleaved and large-cell; Diffuse large cell non-Hodgkin's lymphoma following or concurrent with a diagnosis of follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan; tositumomab I-131

INTERVENTIONS:
Drug: Ibritumomab Tiuxetan
Drug: Iodine I 131 Tositumomab

SUMMARY:
This is a multi-center, randomized, study to compare Iodine I 131 Tositumomab therapeutic regimen to Ibritumomab Tiuxetan therapeutic regimen in the treatment of patients with relapsed or transformed follicular non-Hodgkin's B-cell lymphoma. A total of 350 patients, approximately 175 patients per arm, will be enrolled at 30 to 40 sites in the United States.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis of follicular lymphoma, Grade 1, 2, or 3, or diffuse large cell lymphoma concurrent with or following the diagnosis of follicular lymphoma (WHO/REAL classification).
* International Working Formulation histological equivalents of Follicular, small cleaved; Follicular, mixed small-cleaved and large-cell; follicular large-cell; or Transformed diffuse large cell lymphoma following or concurrent with a diagnosis of follicular lymphoma.
* Patients diagnosed with diffuse large cell lymphoma at study enrollment must have a historical or contemporaneous lymph node biopsy that demonstrates a diagnosis of follicular lymphoma.
* Recurrent lymphoma after at least three qualifying therapy regimens including at least one Rituximab-containing regimen and at least one chemotherapy regimen.
* The patient must have either not responded or responded with a duration of response of less than 6 months to a Rituximab-containing regimen, Performance status of at least 70% on the Karnofsky Scale and an anticipated survival of at least three months.
* Bi-dimensionally measurable disease with at least one lesion measuring 4.0 cm2 by CT scan.
* Absolute neutrophil count >/= 1500 cells/mm3 and platelet count >/=100,000/mm3 within 21 days prior to study enrollment.
* Blood products and/or growth factors should not be taken within 4 weeks prior to blood draw.
* Adequate renal function (defined as serum creatinine <1.5 x upper limit of normal) and adequate hepatic function (defined as total bilirubin <1.5x upper limit of normal and AST <5x upper limit of normal) within 21 days prior to study enrollment.
* Human Anti-Murine Antibody (HAMA) negative within 21 days prior to study enrollment.
* Provision of informed consent as signified by a signed IRB approved consent form prior to any study-specific procedures being implemented.

Exclusion criteria:

* Greater than 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically within 90 days prior to study enrollment.
* Hypocellular bone marrow (</=15% cellularity or marked reduction in bone marrow precursors).
* Prior myeloablative therapy.
* History of failed stem cell collection.
* Prior radiotherapy to fields encompassing more than 25% of the blood forming marrow.
* Prior chemotherapy, biologic therapy, radiation therapy or steroid therapy for NHL within eight weeks prior to screening procedures.
* Prior radioimmunotherapy.
* Prior treatment with any non-human, particularly murine monoclonal or polyclonal antibodies for either diagnostic or therapeutic purposes. This exclusion does not extend to the chimeric monoclonal antibody, Rituximab.
* Prior malignancy other than lymphoma, except for adequately treated basal cell or squamous cell skin cancer, in situ uterine cervical cancer, or other cancer for which the patient has been disease-free for five years.
* Active infection requiring intravenous antibiotics at the time of study enrollment.
* New York Heart Association Class III or IV heart disease or other serious illness that would preclude evaluation.
* HBsAg seropositivity.
* Known HIV infection.
* Known brain or leptomeningeal metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of subjects experiencing Grade 3/4 hematological toxicity within 120 days from completion of treatment regimen administration.

SECONDARY OUTCOMES:
The final analysis will be carried out when 130 events (progressive disease, death or subsequent therapy) have occurred in the control arm, expected approximately 18 months after last subject last visit.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (8):
- United States (8):
  - GSK Clinical Trials Call Center, Iowa City, Iowa
  - GSK Clinical Trial Call Center, St Louis, Missouri
  - GSK Clinical Trials Call Center, Buffalo, New York
  - GSK Clinical Trials Call Center, Charleston, North Carolina
  - GSK Clinical Trial Call Center, Portland, Oregon
  - GSK Clinical Trial Call Center, Knoxville, Tennessee
  - GSK Clinical Trial Call Center, Seattle, Washington
  - GSK Clinical Trials Call Center, Tacoma, Washington